CLINICAL TRIAL: NCT03665324
Title: Atrial Function and Supraventricular Arrhythmia of the Veteran Athlete.
Acronym: FA2V
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3066
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Supraventricular Arrhythmias
Keywords: Supraventricular arrhythmias; veteran athlete; ECG; ETT

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Veteran athletes with Supraventricular arrhythmias: Subjects who consulted in the Sports Medicine Department between January 1, 2010 and January 1, 2017 Veteran athletes (age> 35 years) with documented paroxysmal supraventricular arrhythmias.
  Interventions: Other: Evaluation of the relationship between atrial remodeling evaluated by ECG and ETT with the occurrence of supraventricular arrhythmias
- Veteran athletes without supraventricular arrhythmia: Subjects who consulted in the Sports Medicine Department between January 1, 2010 and January 1, 2017 Veteran athletes (age> 35 years) without documented supraventricular arrhythmia.
  Interventions: Other: Evaluation of the relationship between atrial remodeling evaluated by ECG and ETT with the occurrence of supraventricular arrhythmias

INTERVENTIONS:
Other: Evaluation of the relationship between atrial remodeling evaluated by ECG and ETT with the occurrence of supraventricular arrhythmias — Subjects will be retrospectively retrieved from the Sport Medicine Service of Rennes University Hospital database.
  Medical data will then be collected from the athletes' medical records. The ECG present in the medical file will be reinterpreted to obtain the resting heart rate, the amplitude of the P wave, the morphology of the P wave and the duration of the PR space.
  The data from the stress test will be found from reports in the medical records: resting heart rate, maximum heart rate, sustained peak load, arrhythmia during the test.
  ETTs will be retrieved from the local server. They will be reinterpreted to collect anatomical and functional cardiac data necessary for the study.

SUMMARY:
Supraventricular arrhythmias (including atrial fibrillation) are the most common arrhythmias of the veteran athlete and have a major impact in terms of morbidity and mortality. Although moderate sports practice has been shown to decrease the occurrence of these arrhythmias, it has also been shown that very intense athletic activity is associated with an increased risk of developing atrial fibrillation. The pathophysiological mechanism is not clearly understood. However, it has already been shown that intensive sports practice leads to electrical and morphological atrial remodeling, which could be the cause of the occurrence of supraventricular arrhythmias for these athletes.

For sedentary patients, two major tools predict the risk of the onset of supraventricular arrhythmia: the electrocardiogram (ECG) and transthoracic echocardiography (ETT), particularly with the study of atrial function by the analysis of myocardial deformities.

DETAILED DESCRIPTION:
No studies have tested these two tools for the evaluation of atrial remodeling of the veteran athlete to predict which ones are at risk of developing supraventricular arrhythmias.

However, the identification of predictive factors would make it possible to identify at-risk athletes and thus provide them with adapted sporting practice advice and personalized follow-up.

The aim of the study is to evaluate the relationship between atrial remodeling assessed by ECG and ETT with the occurrence of supraventricular arrhythmia by comparing an athlete group with supraventricular arrhythmia with a control group of healthy athletes.

ELIGIBILITY:
Inclusion Criteria:

* Supraventricular arrhythmia group : Veteran athletes with documented paroxysmal supraventricular arrhythmias.
* Control Group : Veteran athletes without documented supraventricular arrhythmia.

Exclusion Criteria:

* Any cardiopathy (valvulopathy, coronary heart disease, etc.).
* Minor patients,
* Major patients subject to legal protection (legal safeguards, guardianship)
* Persons deprived of their liberty
* Patients opposed to the use of their personal data.

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Veteran athletes who consulted in the Sports Medicine Department between January 1, 2010 and January 1, 2017
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Study of atrial function by analysis of myocardial strain. | At the inclusion day
  Myocardial strain in extracted from ETT and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: frederic SCHNELL, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No